CLINICAL TRIAL: NCT04378647
Title: A Randomized Phase IIb Study, Evaluating Efficacy of Salvage Therapy With Brentuximab Vedotin-ESHAP vs ESHAP in Patients With Relapsed / Refractory Classical Hodgkin's Lymphoma, Followed by Brentuximab Vedotin Consolidation (Instead of Autologous Hematopoietic Stem Cell Transplantation) in Those Who Attained a Metabolic Complete Remission After Salvage Therapy
Brief Title: BREntuximab Vedotin in SEcond LIne Therapy BEfore Transplant
Acronym: BRESELIBET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GELTAMO18-HL
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Hodgkin Lymphoma, Adult
MeSH Terms: conditions — Hodgkin Disease | interventions — Neoadjuvant Therapy; Brentuximab Vedotin; ESAP protocol; Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction ESHAP (Active Comparator): 3 Cycles ESHAP ( 21 days) : Etoposide [40 mg/m2/ day IV, D1-4], Solumedrol [250 mg/day IV, D1-4], High dose Ara-C [2 g/m2 IV, D5] Cisplatinum [25 mg/m2/day IV, D1-4]
  Interventions: Drug: Induction without Brentuximab Vedotin; Drug: Consolidation with Brentuximab Vedotin
- Induction BV-ESHAP (Experimental): 3 Cycles of Brentuximab VEedotin + ESHAP ( 21 days) : Etoposide [40 mg/m2/ day IV, D1-4], Solumedrol [250 mg/day IV, D1-4], High dose Ara-C [2 g/m2 IV, D5] Cisplatinum [25 mg/m2/day IV, D1-4] Brentuximab Vedotin [1.8 mg/kg IV, D1]
  Interventions: Drug: Induction with Brentuximab vedotin (BV); Drug: Consolidation with Brentuximab Vedotin

INTERVENTIONS:
Drug: Induction with Brentuximab vedotin (BV) — 3 cycles ESHAP plus antibody-drug conjugate brentuximab vedotin (BV) at a dose of 1.8 mg/kg IV
  Other Names: Adcetris treatment + ESHAP as salvage therapy
  Arms: Induction BV-ESHAP
Drug: Induction without Brentuximab Vedotin — 3 cycles of ESHAP as a standard of care therapy for those patients with primary refractory cHL and those patients relapsing after first-line therapy
  Other Names: ESHAP treatment as salvage therapy
  Arms: Induction ESHAP
Drug: Consolidation with Brentuximab Vedotin — Up to 13 or 16 cycles of antibody-drug conjugate brentuximab vedotin (BV) at doses of 1.8 mg/kg iv every 21 days)
  Other Names: Adcetris treatment as consolidation

SUMMARY:
A Randomized Phase IIb Study, Evaluating Efficacy of Salvage Therapy with Brentuximab Vedotin-ESHAP vs ESHAP in Patients with Relapsed / Refractory Classical Hodgkin's Lymphoma, Followed by Brentuximab Vedotin Consolidation (instead of Autologous Hematopoietic Stem Cell Transplantation) in Those who Attained a Metabolic Complete Remission after Salvage Therapy

DETAILED DESCRIPTION:
A phase IIb open label multi-center trial in patients with refractory / relapsed cHL.

Patients are randomized (1:1) to receive:

• ESHAP- BV (Etoposide [40 mg/m2/ day IV, D1-4], Solumedrol [250 mg/day IV, D1-4], high dose Ara-C [2 g/m2 IV, D5] and cisplatinum [25 mg/m2/day IV, D1-4] + BV [1.8 mg/kg IV, D1], every 21 days (3 cycles, q21 days).

Or

• ESHAP (Etoposide [40 mg/m2/ day IV, D1-4], Solumedrol [250 mg/day IV, D1-4], high dose Ara-C [2 g/m2 IV, D5] and cisplatinum [25 mg/m2/day IV, D1-4] (3 cycles, q21 days)

Stem cell collection will be performed in all patients according to institutional guidelines, but preferably after the first / second cycle of ESHAP-BV or ESHAP.

Patients attaining a mCR (Deauville 1, 2) after receiving 3 cycles of ESHAP-BV, will receive up to 13 cycles of BV consolidation (administered every 3 weeks, over 39 weeks).

Patients who were randomized to ESHAP and attained a mCR after receiving 3 cycles will receive up to 16 cycles of BV (same dosage and time intervals).

Patients who attained less than mCR following ESHAP-BV/ESHAP they will be taken out of the trial and will be treated according to their physician's clinical decision. However, they will be followed in order to evaluate their clinical outcome in terms of ORR, CR rate, TTNT2 and OS, that will be analyzed the study separately.

ELIGIBILITY:
Inclusion Criteria:

Patients with classical HL CD30+ confirmed histologically (either at the time of diagnosis / at the time of first relapse) will be included in the trial

* Male or female patients 18 to 65 years of age
* Voluntary written informed consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse
* Male patients, even if surgically sterilized, (i.e., status post-vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse
* ECOG 0 to 2
* Measurable disease at time of enrolment (lymphadenopathy/ extranodal mass of at least 1.5 cm)
* No evidence of neuropathy grade ≥2
* Clinical laboratory values as specified in the protocol below within 7 days before the first dose of study drug

Exclusion Criteria:

* Lymphocyte predominant nodular Hodgkin's lymphoma
* Prior treatment with brentuximab vedotin
* Female patient who are both lactating and breast-feeding or have a positive serum pregnancy test during the screening period or a positive pregnancy test on Day 1 before first dose of study drug
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol.
* Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of progressive multifocal leukoencephalopathy (PML)
* Symptomatic neurologic disease compromising normal activities of daily living or requiring medic
* Any sensory or motor peripheral neuropathy greater than or equal to Grade 2
* Known history of any of the following cardiovascular conditions defined in the protocol
* Any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first study drug dose
* Patients that have not completed any prior treatment chemotherapy and/or other investigational agents within at least 5 half-lives (or 28 days if the half-lives are unknown) of last dose of that prior treatment
* Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin.
* Known human immunodeficiency virus (HIV) positive
* Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
* Focal radiation therapy within 30 days prior to study recruitment
* Major surgery within 28 days prior to randomization
* Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have evidence of residual disease.
* Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
PET-CT result | 4-6 weeks after the Cycle 3 started (each cycle is 21 days)
  PET-CT negative, Deauville scores 1 and 2

SECONDARY OUTCOMES:
progression-free survival (PFS) | At the end of two years of last dose of consoldation Brentuximab VEdotin treatment
  Evaluation of patient without progression of disease
Duration of response | At the end of two years of last dose of consoldation Brentuximab VEdotin treatment
  Lenght of time between date of evidence response and progression of disease or death
Overall Survival (OS) | At the end of two years of last dose of consoldation Brentuximab VEdotin treatment
  Time from entry onto the clinical trial (random assignment in a phase III study) until death as a result of any cause.
Duration of response (DOR) | At the end of two years of last dose of consoldation Brentuximab VEdotin treatment
  Time from first documentation of CR or PR to disease progression

OTHER OUTCOMES:
Safety and tolerability | At the end of the 3 years of of last dose of consoldation Brentuximab VEdotin treatment
  AEs, fertility,infections, and secondary malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sureda, PhD, Principal Investigator — Institut Català d'Oncologia, Hospital Duran i Reynals
Locations (19):
- Spain (19):
  - Institut Català D'Oncologia - Hospital Germans Trias I Pujol, Barcelona, Barceolna
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Institut Català D'Oncologia - Hospital Duran I Reynals, Barcelona
  - Institut Català D'Oncologia, Barcelona
  - Hospital Universitario de Cruces, Bilbao
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario J.M. Morales Meseguer, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocío, Seville
  - Hospital Universitario Y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia